CLINICAL TRIAL: NCT04322669
Title: Pidotimod in Children With Recurrent Respiratory Tract Infections (RRI), A Randomized, Double Blind, Placebo Controlled Clinical Trial (P-CRESCENT)
Brief Title: Study of Pidotimod in Children With Recurrent Respiratory Tract Infections (RRI)
Acronym: P-CRESCENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-PIMOT-40
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Respiratory Tract Infections
Keywords: Pidotimod; Recurrent Respiratory Tract Infections; Pediatrics Study
MeSH Terms: conditions — Respiratory Tract Infections | interventions — pidotimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pidotimod (Experimental)
  Interventions: Drug: Pidotimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pidotimod — Participants will be randomized in ratio of 1:1 to receive Pidotimod 400 milligrams (mg), once daily (no infection present) or twice daily (infection present) orally up to Day 60 during the double-blind treatment period.
  Arms: Pidotimod
Drug: Placebo — Participants will be randomized in ratio of 1:1 to receive placebo matched to Pidotimod, once daily (no infection present) or twice daily (infection present) orally up to Day 60 during the double-blind treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of pidotimod as treatment in participants with recurrent respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Participants having the study informed consent signed by their parent(s) / guardian. Participants will also assent specifically for their study participation signing an independent assent form. Site specific ethics requirements will be followed
* Participants with history of respiratory tract infections (Chinese Clinical Concept and management of recurrent respiratory tract infections in children [revised] (2008) (Zhonghua er ke za zhi = Chinese journal of Pediatrics; 46 (2): 108-10) of either:

  * at least the following episodes of upper respiratory tract infections (ear/nose/throat) in the last year: 6 for those aged 3-5 years old at inclusion; 5 for those aged 6-14 years old at inclusion
  * OR at least 2 episodes of lower respiratory tract infections (trachea/bronchia/lungs) in the last 12 months
* Participants compliant with the pidotimod Chinese approved label (package insert) requirements

Exclusion Criteria:

* Participants with any immunodeficiency condition, either primary or secondary (including Acquired immunodeficiency syndrome [AIDS], cancers of the immune system, immune-complex disease, chemotherapy, and radiation)
* Participants with known allergies or hypersensitivity to pidotimod or any of its excipients. Antibiotics allergic participant will not be excluded; but due warning will be given
* Participants with immunomodulatory treatment washout period of less than 4 weeks up to baseline visit
* Participants with any concomitant severe disease at the time of screening that are judged by the investigator that could be detrimental to the participant or could compromise the study (e.g. congenital heart disease, Rheumatic immune disease, congenital deformity of trachea, chronic pulmonary disease, chronic liver and kidney disease, etc)
* Female pregnant or of child bearing potential, for whom the investigator suspects might maintain sexual intercourse, unless she has a negative blood pregnancy test at screening and agrees to use two methods of contraception during the study
* Participants who has previously completed or withdrawn from this study
* Participants with evidence of significant active neuropsychiatric disease, alcohol abuse or drug abuse, in the investigator's opinion
* Participants currently enrolled in, or discontinued within the last 30 days prior to baseline from a clinical study involving an off-label/new use of an investigational drug or device, or concurrently enrolled in a non-observational clinical study or any other type of medical research judged not to be scientifically or medically compatible with this study
* Participants who is unreliable and unwilling to make him/herself available for the duration of the study and who will not abide by the research unit policy and procedure and study restrictions
* Parents/Caregivers without cell phone, tablet or computer availability

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Rate of Respiratory Tract Infection (RI) per Month During Overall Study Period | Baseline (Day 1) up to end of post-treatment follow-up [Day 180/Early Termination (ET)]
  The mean rate of respiratory infection episodes per month during the overall study period will be analyzed and compared between the reported groups.

SECONDARY OUTCOMES:
Rate of Respiratory Tract Infection (RI) per Month During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The mean rate of RI episodes per month during the post-treatment follow-up period will be analyzed.
Rate of Respiratory Tract Infection (RI) per Month During the Double-blind Randomized Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The RI per month during the double-blind randomized treatment period will be assessed.
Number of Days with Respiratory Tract Infections (RI) During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of days with RI during the double-blind treatment period will be assessed.
Number of Days with Respiratory Tract Infections (RI) During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of days with RI during the post-treatment follow-up will be assessed.
Number of Days with Respiratory Tract Infections (RI) During the Overall Study Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of days with RI during the overall period will be assessed.
Number of Antibiotic Use Days During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of antibiotic use days due to any respiratory infection during the double-blind treatment period will be assessed.
Number of Antibiotic Use Days During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of antibiotic use days due to any respiratory infection during the post-treatment follow-up period will be assessed.
Number of Antibiotic Use Days During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of antibiotic use days due to any respiratory infection during the overall period will be assessed.
Number of Antipyretics Use Days During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of antipyretics use days during the double-blind treatment period will be assessed.
Number of Antipyretics Use Days During the Post-Treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of antipyretics use days due to any respiratory infection during the post-treatment follow-up period will be assessed.
  The number of antipyretics use days during the double-blind 60-day treatment period will be assessed.
Number of Antipyretics Use Days During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of antipyretics use days due to any respiratory infection during the overall period will be assessed.
Percentage of Participants Free of Respiratory Tract Infections (RI) During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The percentage of participants free of RI during the double-blind treatment period will be assessed.
Percentage of Participants Free of Respiratory Tract Infections (RI) During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The percentage of participants free of RI during the post-treatment follow-up period will be assessed.
Percentage of Participants Free of Respiratory Tract Infections (RI) During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The percentage of participants free of RI during the overall period will be assessed.
Number of Hospitalization Days During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of hospitalization days due to any respiratory infection during the double-blind treatment period will be assessed.
Number of Hospitalization Days During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of hospitalization days due to any respiratory infections during the post-treatment follow-up period will be assessed.
Number of Hospitalization Days During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of hospitalization days due to any respiratory infections during the overall period will be assessed.
Percentage of Participants with At Least One Hospitalization During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The percentage of participants with at least one hospitalization due to any respiratory infections during the double-blind treatment period will be assessed.
Percentage of Participants with At Least One Hospitalization During the Post-treatment Follow-Up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The percentage of participants with at least one hospitalization due to any respiratory infections during the post-treatment follow-up period will be assessed.
Percentage of Participants with At Least One Hospitalization During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The percentage of participants with at least one hospitalization due to any respiratory infections during the overall period will be assessed.
Number of Wheezing Attack Days During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of wheezing attack days will be observed in terms of two responses: Yes or No, during the double-blind treatment period. An acute wheezing attack is defined as an episode of progressively increasing shortness of breath, cough, wheezing, chest retraction or tightness, or any combination of these symptoms that lasted at least 6 hours with normal results on chest radiographic examinations. In participants with repeated symptoms, attacks are counted separately only if the participant had been without symptoms for at least 1 week between the end of one episode and the beginning of another.
Number of Wheezing Attack Days During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of wheezing attack days will be observed in terms of two responses: Yes or No, during the post-treatment follow-up period. An acute wheezing attack is defined as an episode of progressively increasing shortness of breath, cough, wheezing, chest retraction or tightness, or any combination of these symptoms that lasted at least 6 hours with normal results on chest radiographic examinations. In participants with repeated symptoms, attacks are counted separately only if the participant had been without symptoms for at least 1 week between the end of one episode and the beginning of another.
Number of Wheezing Attack Days During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of wheezing attack days will be observed in terms of two responses: Yes or No, during the during the overall period. An acute wheezing attack is defined as an episode of progressively increasing shortness of breath, cough, wheezing, chest retraction or tightness, or any combination of these symptoms that lasted at least 6 hours with normal results on chest radiographic examinations. In participants with repeated symptoms, attacks are counted separately only if the participant had been without symptoms for at least 1 week between the end of one episode and the beginning of another.
Number of Asthma Days During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  The number of days of asthma attacks will be observed in terms of two responses: Yes or No, recorded in the e-diary, during the double-blind treatment period. Bronchial asthma is a heterogeneous disease characterized by chronic airway inflammation and airway hyperresponsiveness with main clinical manifestations of recurrent wheezing, cough, shortness of breath and chest tightness.
Number of Asthma Days During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  The number of days of asthma attacks will be observed in terms of two responses: Yes or No, recorded in the e-diary, during the post-treatment follow-up period. Bronchial asthma is a heterogeneous disease characterized by chronic airway inflammation and airway hyperresponsiveness with main clinical manifestations of recurrent wheezing, cough, shortness of breath and chest tightness.
Number of Asthma Days During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  The number of days of asthma attacks will be observed in terms of two responses: Yes or No, recorded in the e-diary, during the overall period. Bronchial asthma is a heterogeneous disease characterized by chronic airway inflammation and airway hyperresponsiveness with main clinical manifestations of recurrent wheezing, cough, shortness of breath and chest tightness.
Number of Participants with Adverse Events (AE) During the Double-blind Treatment Period | Baseline (Day 1) up to end of double-blind treatment (Day 60)
  An AE is defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom or disease, temporally associated with the use of a medicinal product, regardless of its nature, intensity, seriousness, or presumed relationship (causality) to the product or experimental procedure used. Participants who experienced any AE will be assessed during the double-blind treatment.
Number of Participants with Adverse Events (AE) During the Post-treatment Follow-up Period | From end of double-blind treatment (Day 60) up to end of post-treatment follow-up (Day 180/ET)
  An AE is defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom or disease, temporally associated with the use of a medicinal product, regardless of its nature, intensity, seriousness, or presumed relationship (causality) to the product or experimental procedure used. Participants who experienced any AE will be assessed during the post-treatment follow- up.
Number of Participants with Adverse Events (AE) During the Overall Period | Baseline (Day 1) up to end of post-treatment follow-up (Day 180/ET)
  An AE is defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom or disease, temporally associated with the use of a medicinal product, regardless of its nature, intensity, seriousness, or presumed relationship (causality) to the product or experimental procedure used. Participants who experienced any AE will be assessed during the overall study.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (16):
- China (16):
  - Investigator Site 01 Children's Hospital Captial Institute of Pediatrics, Beijing
  - Investigator Site 16, Changchun
  - Investigator Site 09, Changde
  - Investigator Site 12, Changsha
  - Investigator Site 07, Guangzhou
  - Investigator Site 10, Guilin
  - Investigator Site 14, Kunming
  - Investigator Site 03, Nanjing
  - Investigator Site 11, Sanya
  - Investigator Site 02, Shanghai
  - Investigator Site 06, Shantou
  - Investigator Site 13, Shaoyang
  - Investigator Site 05, Tianjin
  - Investigator Site 04, Xiamen
  - Investigator Site 08, Yanji
  - Investigator Site 15, Zhengzhou